CLINICAL TRIAL: NCT00508560
Title: Contingency Management for Smoking Cessation Among Veterans With Schizophrenia or Other Psychoses
Brief Title: Contingency Management for Smoking Cessation Among Veterans With Psychotic Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to low recruitment.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUD-Q
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Nicotine Dependence; Psychotic Disorders
Keywords: Contingency management; Smoking cessation; Psychotic disorders; Veterans
MeSH Terms: conditions — Tobacco Use Disorder; Psychotic Disorders; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Experimental
  Interventions: Behavioral: Contingency Management
- Arm 2 (Active Comparator): Active Comparator
  Interventions: Behavioral: Reward

INTERVENTIONS:
Behavioral: Contingency Management — Participants draw from a fishbowl to obtain tokens when they attend a smoking cessation treatment session. The number of draws will be based upon attendance at consecutive sessions. Tokens include messages of encouragement ("Good job!") or VA canteen vouchers of varying monetary value.
  Arms: Arm 1
Behavioral: Reward — Participants receive set reward (VA canteen voucher) for each week of smoking cessation treatment they attend. The value of the reward will not change regardless of attendance at consecutive sessions.
  Arms: Arm 2

SUMMARY:
This study examines the use of contingent incentives to increase attendance at smoking cessation treatment sessions by smokers with schizophrenia and other psychoses who want to quit smoking. We hypothesize that participants randomized to receive contingent rewards for group attendance will attend more treatment sessions than those in the control group.

DETAILED DESCRIPTION:
Schizophrenia and other psychotic disorders are highly prevalent in the VA population and are associated with high rates of smoking. Although smoking cessations approaches that work for non-schizophrenic patients such as behavioral counseling and medications appear to be efficacious for schizophrenic smokers, a major obstacle in providing adequate treatment is poor attendance at treatment sessions. Contingency management has been shown to shape treatment behavior in non-schizophrenic smokers and to shape other behaviors such as cocaine use and exercise in schizophrenics.

The intention of this project is to examine the use of contingent incentives to increase attendance at smoking cessation treatment sessions by smokers with schizophrenia and other psychoses and to compare two different approaches to providing contingent incentives in this context. Subjects in the experimental condition draw from a fishbowl to obtain tokens when they attend a smoking cessation treatment session. The number of draws will be based upon attendance at consecutive sessions. Subjects in the experimental condition receive a set reward that will not change regardless of attendance at consecutive sessions. We hypothesize that the participants in the experimental condition will attend more smoking cessation group therapy sessions than those in the control condition because they will have the possibility, although not the likelihood, to obtain contingent reinforcement of greater value.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be diagnosed with schizophrenia or any other psychotic disorder, bipolar disorder with psychotic features, or major depression with psychotic features according to the electronic medical record.
* Current nicotine use, defined as smoking 5 or more cigarettes/day for at least 16 of the past 30 days prior to study screening.
* Prospective subjects must indicate willingness to attend smoking cessation group therapy.

Exclusion Criteria:

* Imminent risk for suicide or violence.
* Severe psychiatric symptoms or psychosocial instability likely to prevent participation in the study protocol (i.e., attendance at scheduled sessions, ability to read study materials, and/or ability to comprehend interventions).
* Clinically apparent, gross cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of treatment sessions attended | 11 weeks

SECONDARY OUTCOMES:
Reduction in cigarettes per day | 3 and 6 months
7- and 30-day point prevalence abstinence | 3 and 6 months
Continuous abstinence from quit date | 3 and 6 months
Days to relapse from quit date | Up to 6 months
Change in BPRS scores | 3 and 6 months
Change in PHQ-9 scores | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Saxon, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States